CLINICAL TRIAL: NCT07390396
Title: Effect of Adding Extracorporeal Shock Wave Therapy to Exercises in Rotator Cuff Tendinopathy: A Randomized Controlled Trial
Brief Title: Effect of Adding Extracorporeal Shock Wave Therapy to Exercises in Rotator Cuff Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DU-PT-ESWT-RCT-003
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tendinopathy; Shoulder Pain; Supraspinatus Tendinopathy; Shoulder Dysfunction
MeSH Terms: conditions — Shoulder Pain | interventions — Extracorporeal Shockwave Therapy; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups. Group A (Experimental) will receive extracorporeal shock wave therapy (ESWT) in addition to a rotator cuff and scapular stabilization exercise program.
  Group B (Active Comparator) will perform the same exercise program without ESWT.
  Both groups will be treated for 6 weeks, with three exercise sessions per week.
Who Masked: Participant
Masking Description: The study will use a double-blind design. Participants and the outcome assessor will be blinded to the group allocation. The physiotherapist administering ESWT and exercises will not participate in outcome measurements to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal Shock Wave Therapy (ESWT) with Exercise (Experimental): Participants in this group will receive extracorporeal shock wave therapy (ESWT) applied to the supraspinatus tendon once weekly for 6 weeks, in addition to a rotator cuff and scapular stabilization exercise program performed three times per week.
  ESWT will be applied using a focused probe at 1.5 bar pressure, 1500 shocks per session. Exercises will include strengthening and control exercises for rotator cuff and scapular muscles.
  Interventions: Other: Extracorporeal Shock Wave Therapy (ESWT) with Exercise
- Exercise Therapy Only (Active Comparator): Participants in this group will perform the same rotator cuff and scapular stabilization exercise program as the experimental group, without receiving ESWT.
  The exercise program focuses on strengthening, stretching, and neuromuscular control of shoulder and scapular stabilizers, performed three times per week for 6 weeks.
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Extracorporeal Shock Wave Therapy (ESWT) with Exercise — Focused extracorporeal shock wave therapy (ESWT) will be applied to the supraspinatus tendon at 1.5 bar, 1500 shocks per session, once weekly for 6 weeks, in combination with a rotator cuff and scapular stabilization exercise program performed three times weekly.
  This combination is designed to promote tendon healing, improve strength, and reduce shoulder pain.
  Arms: Extracorporeal Shock Wave Therapy (ESWT) with Exercise
Other: Exercise Therapy — A standardized rotator cuff and scapular stabilization exercise program including strengthening, stretching, and control training for the shoulder complex. Exercises are performed three times weekly for 6 weeks under supervision.
  This program serves as the active control for comparison with ESWT + Exercise.
  Arms: Exercise Therapy Only

SUMMARY:
Rotator cuff tendinopathy (RCT) is one of the most common causes of shoulder pain, resulting in functional limitations and reduced quality of life. Exercise therapy is considered a first-line treatment; however, adjunct modalities such as extracorporeal shock wave therapy (ESWT) may enhance recovery. This study aims to evaluate the effect of adding ESWT to a rotator cuff and scapular stabilization exercise program in patients with rotator cuff tendinopathy.

DETAILED DESCRIPTION:
Rotator cuff tendinopathy involves chronic overload and microtrauma of the rotator cuff tendons, leading to pain, inflammation, and functional impairment. Therapeutic exercises that target the rotator cuff and scapular stabilizers are commonly prescribed to restore muscle control and shoulder kinematics.

Extracorporeal shock wave therapy (ESWT) has demonstrated potential for tendon regeneration, pain reduction, and improved vascularization. This randomized controlled trial investigates whether the combination of ESWT and exercise therapy produces greater improvements than exercise therapy alone in reducing supraspinatus tendon thickness and pain and improving shoulder function.

Fifty participants aged 30-55 years with confirmed RCT will be randomly assigned into two groups:

* Group A (Experimental): ESWT + rotator cuff and scapular stabilization exercises.
* Group B (Active Comparator): Rotator cuff and scapular stabilization exercises only.

Both groups will be treated for 6 weeks, with 3 exercise sessions per week; Group A will receive 1 ESWT session weekly in addition to exercises.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable individuals who consent to participate in the study.
* Male and female participants aged between 30 and 55 years.
* Diagnosed with rotator cuff tendinopathy, confirmed clinically and by ultrasound or MRI.
* Duration of symptoms greater than 3 months.
* Supraspinatus tendon thickness > 5.85 mm as measured by ultrasound (based on Hunter et al., 2021).
* Able to follow the treatment plan and attend all therapy sessions.

Exclusion Criteria:

* Massive rotator cuff tear or complete tendon rupture.
* Adhesive capsulitis or significant limitation of passive shoulder motion.
* History of shoulder fracture, dislocation, or surgery in the affected limb.
* Rheumatoid arthritis, diabetes mellitus, or systemic inflammatory disease.
* Cervical radiculopathy or neurological involvement affecting the shoulder.
* Corticosteroid injection in the affected shoulder within the last 6 months.
* Pregnancy or breastfeeding.
* BMI > 30 kg/m² (obese individuals excluded).
* Current malignancy, open wounds, or local infection at the treatment site.
* Inability to tolerate shock wave therapy or perform exercise sessions.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Supraspinatus Tendon Thickness | Baseline and at 6 weeks post-intervention
  Supraspinatus tendon thickness will be measured using diagnostic ultrasonography in the transverse plane. Participants will be positioned in the modified Crass position (palm on iliac crest, elbow directed posteriorly) as described by Ferri et al. (2005). The transducer will be placed on the acromion and moved laterally to visualize the supraspinatus tendon. A decrease in tendon thickness after 6 weeks of treatment indicates structural improvement. Measurements will be taken at baseline and at 6 weeks post-intervention.
Change in Shoulder Pain Intensity (Numeric Pain Rating Scale, NPRS) | Baseline and at 6 weeks post-intervention
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will rate their average shoulder pain over the previous week. A lower score after treatment indicates improvement. Measurements will be taken at baseline and at 6 weeks post-intervention.
Change in Shoulder Disability (Shoulder Pain and Disability Index, SPADI) | Baseline and at 6 weeks post-intervention
  Shoulder pain and disability will be assessed using the Shoulder Pain and Disability Index (SPADI). This self-reported questionnaire includes 13 items scored from 0-10. The total score is expressed as a percentage, with higher scores indicating greater pain and disability. The SPADI will be administered at baseline and at 6 weeks post-intervention.
Change in Isometric Shoulder Muscle Strength | Baseline and at 6 weeks post-intervention
  Isometric strength of the shoulder external and internal rotator muscles will be measured using a handheld dynamometer. Participants will perform maximal voluntary contractions in a standardized seated position. Three trials will be performed for each direction of movement, and the mean value will be recorded in Newtons (N). Increased strength after treatment indicates functional improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Deraya University, Minya, Menia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michener, L. A., Subasi Yesilyaprak, S. S., Seitz, A. L., Timmons, M. K., & Walsworth, M. K. (2015). Supraspinatus tendon and subacromial space parameters measured on ultrasonographic imaging in subacromial impingement syndrome. Knee Surgery, Sports Traumatology, Arthroscopy, 23(2), 363-369.
- [Background] Lyng, K. D., Andersen, J. D., Jensen, S. L., Olesen, J. L., Arendt-Nielsen, L., Madsen, N. K., & Petersen, K. K. (2022, Oct). The influence of exercise on clinical pain and pain mechanisms in patients with subacromial pain syndrome. Eur J Pain, 26(9), 1882-1895. https://doi.org/10.1002/ejp.2010
- [Background] Liaghat, B., Skou, S. T., Jørgensen, U., Sondergaard, J., Søgaard, K., & Juul-Kristensen, B. (2020). Heavy shoulder strengthening exercise in people with hypermobility spectrum disorder (HSD) and long-lasting shoulder symptoms: a feasibility study. Pilot Feasibility Stud, 6, 97. https://doi.org/10.1186/s40814-020-00632-y
- [Background] Belley, A. F., Gagnon, D. H., Routhier, F., & Roy, J.-S. (2017). Ultrasonographic measures of the acromiohumeral distance and supraspinatus tendon thickness in manual wheelchair users with spinal cord injury. Archives of physical medicine and rehabilitation, 98(3), 517-524.
- [Background] Beshay, N., Lam, P. H., & Murrell, G. A. C. (2011). Assessing the Reliability of Shoulder Strength Measurement: Hand-Held versus Fixed Dynamometry. Shoulder & Elbow, 3(4), 244-251. https://doi.org/10.1111/j.1758-5740.2011.00137.x
- [Background] Fraenkel, L., Cunningham, M., Peters, E., & Seligman, C. (2012). Measuring pain impact versus pain severity using a numeric rating scale. Journal of General Internal Medicine, 27(5), 555-560. https://doi.org/10.1007/s11606-011-1932-1
- [Background] Alsanawi, H. A., Alghadir, A., Anwer, S., Roach, K. E., & Alawaji, A. (2015). Cross-cultural adaptation and psychometric properties of an Arabic version of the Shoulder Pain and Disability Index. International Journal of Rehabilitation Research, 38(3), 270-275. https://doi.org/10.1097/mrr.0000000000000118
- [Background] Breckenridge, J. D., & McAuley, J. H. (2011). Shoulder Pain and Disability Index (SPADI). J Physiother, 57(3), 197. https://doi.org/10.1016/s1836-9553(11)70045-5
- [Background] Xue, X., Song, Q., Yang, X., Kuati, A., Fu, H., Liu, Y., & Cui, G. (2024, May 4). Effect of extracorporeal shockwave therapy for rotator cuff tendinopathy: a systematic review and meta-analysis. BMC Musculoskelet Disord, 25(1), 357. https://doi.org/10.1186/s12891-024-07445-7
- [Background] Wang, X., Jia, S., Cui, J., Xue, X., & Tian, Z. (2024, Sep 18). Effect of extracorporeal shock wave combined with autologous platelet-rich plasma injection on rotator cuff calcific tendinitis: study protocol for a randomized controlled trial. Trials, 25(1), 616. https://doi.org/10.1186/s13063-024-08407-z
- [Background] Fatima, A., Ahmad, A., Gilani, S. A., Darain, H., Kazmi, S., & Hanif, K. (2022). Effects of High-Energy Extracorporeal Shockwave Therapy on Pain, Functional Disability, Quality of Life, and Ultrasonographic Changes in Patients with Calcified Rotator Cuff Tendinopathy. Biomed Res Int, 2022, 1230857. https://doi.org/10.1155/2022/1230857